CLINICAL TRIAL: NCT02997488
Title: Comparison of Routine Endotracheal Intubation With McGrath Videolaryngoscope and Pentax AirwayScope
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiyoung Lee, Clinical assistant prefessor, Ajou University School of Medicine
Other Study IDs: AJIRB-DEV-OBS-16-473
Record Dates: First submitted 2016-12-14; First posted 2016-12-20 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Intubation
Keywords: videolaryngoscope

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- McGrath: McGrath Videolaryngoscope
  Interventions: Device: McGrath Videolaryngoscope
- Pentax: Pentax Airwayscope
  Interventions: Device: Pentax Airwayscope

INTERVENTIONS:
Device: Pentax Airwayscope — intubation using Pentax Airwayscope
  Groups: Pentax
Device: McGrath Videolaryngoscope — intubation using McGrath Videolaryngoscope
  Groups: McGrath

SUMMARY:
Recently many kinds of indirect videolaryngoscopes were developed. These videolaryngoscopes provide easier intubation, help intubation difficulty, are used good tool for education. McGrath Videolaryngoscope and Pentax AirwayScope are kinds of these videolaryngoscopes.

The purpose of this study is to compare of routine endotracheal intubation with McGrath Videolaryngoscope and Pentax AirwayScope by means of providing better laryngeal view, easier and faster intubation.

ELIGIBILITY:
Inclusion Criteria:

* an American Society of Anesthesiologists physical status (ASA) 1 or 2

Exclusion Criteria:

* a suspected difficult airway (Mallampati score Ⅳ)
* known cervical spine injury
* required rapid sequence induction
* emergency operation

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for elective surgery requiring orotracheal intubation in our hospital
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Time to intubation | 10 minutes around intubation
  from entering of blade between incisors to appearance of first end tidal CO2 curve using capnograph

CONTACTS AND LOCATIONS:
Overall Officials: Jiyoung Lee, MD, Principal Investigator — Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No